CLINICAL TRIAL: NCT04438499
Title: e۰Sense® Clinical Investigation: Assessing the Performance, Safety and Usability of e۰Sense® Electronic Catheters for Performing Urodynamic Studies
Brief Title: e۰Sense® Catheter Clinical Investigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laborie Medical Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ESNS-PH01
Record Dates: First submitted 2020-06-02; First posted 2020-06-18 (Actual); Results first posted 2022-09-07 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Urodynamics
Keywords: urodynamics; urinary catheter

STUDY DESIGN:
Intervention Model Description: There will be no control arm or blinding in this trial or inclusion of a sham or placebo, as it is not applicable to the study design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects Indicated for a UDS study (Experimental): The investigational device, i.e. the eSense catheter will be used in all the subjects to assess primary and exploratory objectives. It is a single arm study with no comparative, placebo, sham or control arm.
  Interventions: Device: eSense 7fr Single Sensor Bladder Catheter

INTERVENTIONS:
Device: eSense 7fr Single Sensor Bladder Catheter — Urinary and abdominal catheters inserted in to the body to measure pressure for urodynamics.
  Other Names: eSense 7Fr Abdominal Catheters; eSense 7Fr Dual Sensor Urethral Catheters

SUMMARY:
This pre-market study will be conducted on consenting patients undergoing a medically prescribed, invasive, conventional urodynamics (UDS) test using the investigational device (e۰Sense® urodynamic catheters). Data pertaining to the safety, effectiveness and usability of the catheters will be collected.

DETAILED DESCRIPTION:
The study will recruit and consent up to 65 subjects from up to 4 different sites (minimum 15 subjects recruited at each site) in the European Union, and the expected duration of each subject's participation is one clinic visit to receive their already requested UDS test. A follow-up call will be conducted three to five days later to collect adverse event information post-test. An interim analysis is to be performed when data from 30 patients has been completed to support the primary objective, and using the results for regulatory purposes (e.g. CE marking). However, the study enrollment continues, during the interim analysis, until 60 patients (maximum 65) have been recruited and all data collected. At the end of the study, the data will be analysed against secondary and exploratory objectives including an exploratory analysis of the primary objective on all patients.

To collect data for the study, Case Report Forms (CRF) have been developed. They will be paper based and do not include any patient identifiers except a Site Subject ID. Any document linking the Site Subject ID to subject information will be stored at the site and not shared with the sponsor. Additionally, CRF completion guidelines will be developed prior to study initiation to aid correct and consistent data collection. These guidelines will be provided to the site and site personnel will be trained prior to subject enrollment. CRFs will be treated as source data in the event that the original information is entered on the CRFs first, and no source document worksheet is utilized for that data point. Laborie will enter CRF data in to an excel database that has been developed to represent each field on the CRF. Data Management activities are conducted in accordance with Laborie's Data Management Plan, including but not limited to: source data verification (monitoring), query handling and resolution, data entry quality control and controlled database locking. Guidelines have also been created that contain detailed descriptions of each data entry point and how to enter in the database.

The data from the CRFs will be used to make the following assessments:

* The investigator will be asked to make an assessment to determine the safety and performance of the device regarding the intended use.
* A Numeric Pain Rating Scale (NPRS) will be used to assess the parameters of patient discomfort/pain, if appropriate.
* All adverse events will be recorded to assess the safety of the device.
* Subjective questionnaire completed by the user to assess ease of use, ease of insertion and removal, ease of securing the catheter, tracing stability (overall, during filling, voiding and UPP where applicable), tracing quality (overall, Pves, Pabd, Pura where applicable), channel subtraction quality, visibility on Video Urodynamics (VUDS, where applicable), catheter stiffness, sensor location, patient tolerance, and overall usability performance.
* Pre-test at various positions and resting pressures through the study
* The de-identified urodynamic data files will be collected and stored

Risks to the patient will be no greater than those of a standard Urodynamics test. Patients may experience temporary discomfort upon insertion of the catheters. Test duration may be slightly longer than a standard test while assessment of the study materials is being made, and so discomfort and inconvenience associated with an extended test duration may occur. Furthermore, bladder catheterization can increase the risk of urinary tract infection, but with no higher incidence than during standard urodynamics. No patient follow-up visit is scheduled for this study, unless deemed necessary by the physician in the event of adverse event(s).

Monitors are appointed by Laborie and are appropriately trained with scientific and/or clinical knowledge needed to monitor the trial adequately. The monitors are also thoroughly familiar with the investigational medical device under investigation, the protocol, written informed consent form (ICF), and any other written information to be provided to subjects, Laborie standard operating procedures, ISO 14155, and GCP.

The monitor conducts activities per Laborie's Monitoring Plan, including but not limited to:

* Acting as the main line of communication between the sponsor and the investigator.
* Verifying that the investigator has adequate qualifications, number of subjects, and resources and remain adequate throughout the trial period, and that facilities are adequate to safely and properly conduct the trial and remain adequate through the trial period.
* Initiating each participating sites
* Ensuring the investigational device is being used according to the protocol and instructions for use
* Verifying that the investigator and investigation site team understands and follows the approved protocol and all approved amendments (if any).
* Verifying that the investigator is familiar with the responsibilities of the principal investigator.
* Ensuring the investigator and site team are informed and knowledgeable of all relevant document updates concerning the clinical trial.
* Ensuring that the investigator receives the most up-to-date copy of the Investigator's Brochure, all documents, and all trial supplies needed to conduct the trial properly and to comply with the applicable regulatory requirements.
* Verifying that only authorized and trained site personnel are participating in the clinical trial.
* Verifying that source data and other records are accurate, complete, up to date, stored, and maintained appropriately.
* Signed and dated informed consent forms have been obtained from each subject at the point of enrolment or before any clinical-investigation-related procedures are performed.
* Verifying that CRFs and queries are complete, recorded in a timely manner, and consistent with SD.
* Verifying that appropriate corrections, additions, or deletions are made to the CRFs, dated, explained if necessary and initiated by the authorized designee. The monitor shall NOT make corrections, additions, or deletions to the CRFs.
* Ensuring all adverse events (AEs) and device deficiencies (DDs) are reported to the sponsor and all serious AEs as well as DDs that could have led to serious adverse device events are reported to the sponsor without unjustified delay.
* Verifying that subject withdrawal has been documented and that subject or site non-compliance with the requirements has been documented.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female subjects (Age: 21 years and over) who are medically indicated for UDS testing.

Exclusion Criteria:

* Subjects with significant cognitive deficiency that prevent the subject from giving informed consent
* Subjects suffering from an active bladder infection (not including subjects with asymptomatic bacteriuria)
* Pregnant women
* Subjects with recent (less than 2 weeks) pelvic floor surgery
* Subjects who require the use of a suprapubic catheter

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2023-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Kirschner-Hermanns, MD, Principal Investigator — Rehabilitationszentrum Godeshöhe; Gérard Amarenco, Prof, M.D., Principal Investigator — Hôpital Tenon AP-HP, Sorbonne Université
Locations (2):
- Hôpital Tenon AP-HP (Sorbonne Université), Paris, France
- Rehabilitationszentrum Godeshöhe, Bonn, Germany

REFERENCES:
- [Background] Fleiss, J.L., Levin, B., & Cho Paik, M. (2003). Statistical Methods for Rates and Proportions (3rd ed.). New York, NY: Wiley

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects Medically Indicated for a Urodynamics (UDS) Study: The investigational device, i.e. the eSense catheter will be used in all the subjects to assess primary and exploratory objectives. It is a single arm study with no comparative, placebo, sham or control arm.
  eSense 7fr Catheters: A bladder and abdominal catheter are inserted in to the body to measure pressure for urodynamics.
Period: Overall Study
Arm/Group | Subjects Medically Indicated for a Urodynamics (UDS) Study
Started | 61 (Final sensitivity analysis population)
Completed | 58
Not Completed | 3
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Population: All eligible subjects medically indicated for a urodynamics (UDS) study are included in the baseline analysis population.
Arm/Group | Subjects Medically Indicated for a Urodynamics (UDS) Study
Number analyzed (Participants) | 61
Age, Continuous [Mean (Full Range); unit: years] | 53.9 [31 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 30
  France | 31

OUTCOME MEASURES:

1. Primary Outcome: Clinician Safety and Effectiveness Rating of eSense Catheters (Per Patient)
Description: The primary objective of the study is to gather clinical data to confirm that the updated e۰Sense® catheters are safe and effective for urodynamic use in subjects medically indicated for urodynamics testing.
  The primary outcome will be measured by recording the clinician safety and effectiveness rating for each subject on their CRF. The clinicians will indicate whether each of the e۰Sense® bladder and abdominal catheters are safe & effective for urodynamic use. Given the intended use of the device, and the fact that there is no single or combined objective measures generated from the UDS test that can establish the safety and effectiveness, it is justified to obtain clinicians' feedback via a binary response whether the device is safe and effective for urodynamic use.
Time Frame: approximately 60 minutes
Population: Sensitivity analysis "Intent to treat" population.
Measure: Count of Participants; unit: Participants
Groups:
- Subjects Medically Indicated for a UDS Study: The investigational device, i.e. the eSense catheter will be used in all the subjects to assess primary and exploratory objectives. It is a single arm study with no comparative, placebo, sham or control arm.
  eSense 7fr Single Sensor Bladder Catheter: Urinary and abdominal catheters inserted in to the body to measure pressure for urodynamics.
Arm/Group | Subjects Medically Indicated for a UDS Study
Number analyzed (Participants) | 61
Participants | 58

2. Secondary Outcome: To Report the Percentage of Participants Free From Severe Complication for the Updated e۰Sense Catheters
Description: The secondary outcome will be measured by recording the percentage of participants that do not experience a severe complication or a serious adverse event (as defined in the protocol). Due to the low risk profile of UDS, the sponsor would like to report the severe complication-free rate for any severe complications associated with UDS, and therefore this secondary safety endpoint was planned. Additionally, the sponsor would like to collect and assess this information due to a lack of available published data using the e۰Sense® catheter technology.
Time Frame: approximately 60 minutes
Population: sensitivity analysis population
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Received a Urodynamics Test Using eSense Catheters Free From Severe Complication: The number of participants analyzed for this outcome measure represents the number and percentage of participants free from severe complication who received a urodynamics test using eSense catheters.
Arm/Group | Participants Who Received a Urodynamics Test Using eSense Catheters Free From Severe Complication
Number analyzed (Participants) | 61
Participants | 61

3. Other Pre Specified Outcome: Assess User Impression Based on Subjective Measures
Description: Assess user impressions of the updated e۰Sense® catheters compared with their experience using the existing catheters at each site, by evaluating the following subjective measures: ease of use, ease of insertion and removal, ease of securing the catheter, tracing stability, tracing quality , channel subtraction quality, visibility on VUDS (where applicable), catheter stiffness, sensor location, subject tolerance, and overall usability performance.
  This exploratory endpoint will be measured by collecting usability data in a questionnaire format. At the end of each clinic day a trained clinical user shall complete the questionnaire. When evaluating the usability of a device, the sponsor feels it's appropriate to use a subjective ordinal scale response while assessing human and device usability factors.
Time Frame: approximately 60 minutes
Reporting Status: Not Posted, anticipated posting 2024-10

4. Other Pre Specified Outcome: Asses Subjective Discomfort Levels in the Study Population
Description: Outcome not included in a priori interim analysis plan as per the protocol. Assess subjective subject feedback regarding their discomfort and pain levels. This exploratory endpoint will be measured by collecting subject feedback regarding the level of discomfort and pain experienced during their Urodynamic test using the Numerical Pain Rating Scale (NPRS). Subjects will grade their discomfort/pain on the NPRS from 0 ("No Pain") to 10 ("Worst Pain"). Given the subject population, use of the NPRS is a validated tool in evaluating pain ratings in adults.
Time Frame: approximately 60 minutes
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Assess Resting Pressures in the Subject Before Urodynamics
Description: Outcome not included in a priori interim analysis plan as per the protocol. This exploratory endpoint will be measured by recording initial resting pressures (in cmH20) using the updated e۰Sense® catheters while each subject is positioned in a sitting, standing and supine position, if patient mobility allows. Resting pressures will be recorded on each subjects' CRF 1 during their urodynamics visit.
Time Frame: approximately 60 minutes
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Assess Resting Pressure at Different Filling and Emptying Volumes
Description: Outcome not included in a priori interim analysis plan as per the protocol. This exploratory endpoint will be measured by recording resting pressures (in cmH20) using the updated e۰Sense® catheters during various points of the UDS test as applicable (every 100 mL of filling, MCC, and post-void) at the recorded patient position (sitting, standing, or supine). Patients are to remain in the same position throughout, however supplemental positions can be used (e.g. performing provocative manoeuvres). Resting pressures and patient position will be recorded on each subjects' CRF 1 during their urodynamics visit.
Time Frame: approximately 60 minutes
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The duration of each patient's participation was one clinic visit with a follow-up call 3-5 days later, after which their involvement in the study ended.
Description: Referencing the Medical Device Safety Plan Ordinance (MPSV) under German law:
  Serious Adverse Event - MPSV § 2 (5) English: A serious adverse event (SAE) is any undesired event occurring in a clinical investigation or a performance evaluation study requiring an authorization, which has led, or could have led, or could lead directly or indirectly to the death or severe health impairment of volunteers, users or other persons regardless of whether the event was caused by the medical device.
Arm/Group | Subjects Medically Indicated for a Urodynamics (UDS) Study
All-Cause Mortality (participants affected / at risk) | 0/61
Serious Adverse Events (participants affected / at risk) | 0/61
Other Adverse Events (participants affected / at risk) | 13/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Medically Indicated for a Urodynamics (UDS) Study (N=61)
Mild discomfort in the urethra (Renal and urinary disorders) | 10 (10) — Mild discomfort in the urethra following catheterization that was short lasting and resolved without intervention.
Mild macrohematuria (Renal and urinary disorders) | 3 (3) — Small amount of blood when passing urine.
Diarrhea (Gastrointestinal disorders) | 1 (1)
Bleeding upon catheter removal (Renal and urinary disorders) | 1 (1) — Mild bleeding upon removal of vesical (bladder) catheter

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-24): https://cdn.clinicaltrials.gov/large-docs/99/NCT04438499/Prot_SAP_000.pdf